CLINICAL TRIAL: NCT02248363
Title: Nationwide Evaluation of Multimodal Rehabilitation in Patients With Chronic Musculoskeletal Pain: Treatment Effectiveness and Prediction
Brief Title: Nationwide Evaluation of Multimodal Rehabilitation in Patients With Chronic Musculoskeletal Pain
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Karolinska Institutet (Other)
Collaborators: The Swedish Research Council (Other Government); Karolinska Institutet: Doctoral School in Health Care Sciences (NFV) (Unknown)
Responsible Party: Principal Investigator, Björn O. Äng, Associate professor, Karolinska Institutet
Other Study IDs: Chronic-pain-effect-prediction
Record Dates: First submitted 2014-09-21; First posted 2014-09-25 (Estimated); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Chronic Pain; Widespread Chronic Pain
Keywords: Rehabilitation; Effectiveness; Determinants; Prediction
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Multimodal rehabilitation — Multimodal rehabilitation (MMR) distinguishes itself as an interdisciplinary-coordinated (e.g., physician, occupational therapist, physiotherapist, and psychologist) intervention using a bio-psycho-social view of chronic pain. The MMR continues over a lengthy period with a common goal and generally includes patient education, supervised physical activity, simulated work training, and cognitive behavioural therapy (CBT). The exact composition of these MMR components depends on initial evaluations of the patients health status and furhter follow-up testing. The MMR interventional components can act independently and interdependently, resulting in combined effects due to known and unknown mechanisms; the effects are intended to be greater than the sum of its components.
  Other Names: Multidiciplinary rehabilitation

SUMMARY:
Chronic pain is a common health problem that causes enormous social costs. A common method for treating patients with chronic pain problems are multimodal rehabilitation (MMR), which consists of a combination of physical exercise, cognitive behavioural therapy and work training coordinated in an interdisciplinary team. Our research aims to evaluate the effectiveness of MMR on health, quality of life, physical activity, return to work and health economics, with the long-term goal of developing MMR. We aim also to evaluate predictive factors for good and bad treatment outcomes in order to better adapt the MMR to the patient. The project is based on patient-reported data from the Swedish Quality Registry for Pain Rehabilitation, which routinely collects data from 40 (2017) Swedish specialist MMR clinics from all parts of the country. We expect increased knowledge of treatment effects and how MMR can be effectively adapted according to the patient's limitations and resources. Our project group is interdisciplinary and is active in nationwide research networks that focus on chronic pain and rehabilitation.

DETAILED DESCRIPTION:
Chronic musculoskeletal pain is a public health problem, which frequently cause long-term sickness absence (>180 days). Societal costs of chronic pain are immense, with direct and indirect costs amounting to 90 billion Swedish crowns per year according to Swedish Council on Technology Assessment (SBU). Despite this, few policies have aimed specifically at chronic pain as a public health problem, also acknowledged in the later literature. Multimodal rehabilitation (MMR) is an increasingly used method in this patient group and denotes a combination of psychological measures, physical activity/exercise and manual or physical methods, administered by multidisciplinary teams. Its approach considers the patient's needs from a bio-psycho-social perspective, including work or employment status. At date, MMR is commonly offered by a number of specialist clinics throughout Sweden, of which more than 95% (currently 40) are connected to the Swedish Quality Registry for Pain Rehabilitation (SQRP) with the purpose to collect data for work with quality improvement and research.

According to the latest report from SBU, medium to high evidence from available research supports that MMR is effective for patients with chronic pain, with a few studies suggesting that MMR is superior to traditional and single-treatment programs. However, there is a paucity in the scientific literature with respect to how MMR should be designed to optimize results, and comparisons between different MMR designs or durations are limited. This void is a cause for uncertainty which delays improvement of existing MMR programs treating patients with chronic pain. Further, it is necessary to investigate whether reported results from RCTs and systematic reviews truly apply to naturalistic practice settings with a consecutive non-selective flow of patients, which may be done using a research methodology known as practice-based evidence through prospective observational cohort study designs. Our intention with the present research program is therefore to clarify effectiveness of different MMR designs. Furthermore, knowledge on risk predictors of poor treatment outcomes, and how long-term pain can be prevented and treated is greatly limited. Here, it is currently unclear what factor, patient related and/or treatment component, are more or less effective in different subgroups of patients with chronic pain. This has been discussed in the national SQRP-network and is in demand in the scientific literature. Knowledge of this will enable MMR providers to customize treatment according to patient profile in order to maximize treatment outcomes in relation to costs.

The overall aim of this research program is to prospectively evaluate multimodal rehabilitation (MMR) in patients with chronic pain conditions. The long-term goal is to develop and implement updated knowledge into Swedish MMR programs. The following two strategic aims will be targeted: 1) effectiveness of MMR programs with different durations (short, moderate and long-duration) , 2) prediction and risk of positive and negative outcomes, respectively.

Methods Study design This research project is carried out with longitudinal cohort-study designs based on data extracted from the Swedish Quality Registry for Pain Rehabilitation (SQRP; www.ucr.uu.se/nrs). Data covering several years will be used to analyse the effects of MMR. We expect a large sample size, it entail high test-power for the analyses of overall effects. Therefore, in addition to tests of statistical significance, effect sizes will be calculated in order to avoid type I error, i.e. avoid to falsely claiming that effect exists with support the support of p-values in such large sample. Included subjects are patients aged between 16 and 67 with a referral to a MMR clinic (specialist clinic) for chronic musculoskeletal pain problems.

Data from SQRP allows for longitudinal evaluation of treatment effects, prediction analyses. SQRP is a registry mainly covering patient-reported questionnaire data intended for health care research and quality work for healthcare providers that offer MMR. SQRP is connected to the Swedish Association of Local Authorities and Regions (Sveriges Kommuner och Landsting) and part of a system of national quality registries in Sweden (www.kvalitetsregister.se). Currently, 40 Swedish MMR specialist-treatment units (representing over 95% of the pain rehabilitation centres in the country) are associated with the registry and continuously transmit their patient data to SQRP (www.ucr.uu.se/nrs/index.php/om-registret). This means that nationwide data from all parts of Sweden is included in SQRP which constitutes a major strength of this database. Based on this data, an annual report is compiled by the SQRP steering group and co-workers describing and comparing the performance of the associated MMR treatment units on the overall scale. Since 2007 these accounts have been available to the public (http://www.ucr.uu.se/nrs/index.php).

Data from established questionnaires are registered in SQRP to measure health-related quality of life (SF-36), the consequences of prolonged pain problems on the level of activity and function (Multidimensional Pain Inventory, MPI), perceived health (EQ-5D), pain intensity (numeric rating scale), and anxiety and depression (The Hospital Anxiety and Depression Scale, HAD). Furthermore, data on socio-demographic details, information on employment and sick leave status as well as pain duration and future prospects is collected. In addition to the patient-reported data, an attending MMR practitioner complements the registry with the patient's diagnosis, information on type of pain and expected form of employment (post-rehabilitation).

Data analysis Health-related quality of life, pain intensity, function, activity level, as well as anxiety will serve as dependent outcome measures in the evaluation of effects. The use of a single outcome measure is rarely sufficient to describe the patient's experience, symptoms or treatment outcome in terms of understanding potential effects. However, multiple outcome variables can be inter-correlated and therefore it is reasonable to apply multivariate analyses to control for such dependent relationships. Therefore, multivariate repeated measures analyses will be used to approach effect variables prospectively, while logistic regressions (or similar) with a multiple approach will be applied to analyse prediction models.

ELIGIBILITY:
Inclusion Criteria:

* Chronic pain, e.g. long-term neck and back pain or progressed generalized widespread pain that has lasted more than three months
* 18 to 67 yrs old
* Referred to one of the specialist MMR-clinical department in Sweden

Exclusion Criteria:

- Malignancies

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Included subjects are patients with chronic pain conditions not caused by malignancies (mainly musculoskeletal pain) aged between 18 and 67.
Sampling Method: Probability Sample
Enrollment: 6500 (Estimated)
Dates: Start 2014-09; Primary Completion 2020-10-31 (Estimated); Study Completion 2020-10-31 (Estimated)

PRIMARY OUTCOMES:
Health-related quality of life (SF-36) | Change from baseline to post-treatment, and at 12 months follow-up.
  The SF-36 is a self-assessed multi-purpose, short-form health survey with only 36 questions. It yields an 8-scale profile of functional health and well-being scores as well as psychometrically-based physical and mental health summary measures and a preference-based health utility index. It is a generic measure, as opposed to one that targets a specific age, disease, or treatment group. Accordingly, the SF-36 has proven useful in surveys of general and specific populations, comparing the relative burden of diseases, and in differentiating the health benefits produced by a wide range of different treatments.

SECONDARY OUTCOMES:
Multidimensional Pain Inventory (MPI) | Change from baseline to post-treatment, and at 12 months follow-up.
  The Multidimensional Pain Inventory (MPI) is a self-assessed comprehensive instrument for assessing a number of dimensions of the chronic pain experience, including pain intensity, emotional distress, cognitive and functional adaptation, and social support. It is one of the best instruments available for assessing overall adjustment of chronic pain patients and the outcomes of treatment interventions.
Perceived health (EQ-5D) | Change from baseline to post-treatment, and at 12 months follow-up.
  EQ-5D is a self-assessed standardised measure of health status. It provides a simple, generic measure of health for clinical and economic appraisal. It is applicable to a wide range of health conditions and treatments, it provides a simple descriptive profile and a single index value for health status that can be used in the clinical and economic evaluation of health care as well as in population health surveys.
Pain intensity (numeric rating scale, NRS) | Change from baseline to post-treatment, and at 12 months follow-up.
  The Numeric Rating Scale is a simple reporting instrument that can help to quantify a patient's subjective pain. The Numeric Rating Scale is administered by asking the patient to verbally estimate his or her pain on a scale of 0 to 10, with 0 representing no pain and 10 representing the worst possible pain.
The Hospital Anxiety and Depression Scale, HAD | Change from baseline to post-treatment, and at 12 months follow-up.
  The Hospital Anxiety and Depression Scale (HAD) is a widely used patient self-rated scale with 14 questions (7 "anxiety" and 7 "depression" questions) that ranges from 0-42. It is a well-documented instrument for assessing symptoms of anxiety and depression in patients with somatic diseases.

CONTACTS AND LOCATIONS:
Overall Officials: Björn Äng, Assoc prof., Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Huddinge, Stockholm County, Sweden